CLINICAL TRIAL: NCT03972020
Title: Mindful-life: a Randomized Clinical Trial to Evaluate the Efficacy of a Mindfulness Based Intervention as Compared to Cognitive Behavioral Therapy for Depressive Symptoms and Quality of Life in Patients With Breast Cancer
Brief Title: Mindful-life: Mindfulness Based Intervention vs Cognitive Behavioral Therapy in Patients With Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, luca ostacoli, Associate professor of clinical psychology, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OstacoliMIND&BC
Record Dates: First submitted 2019-02-11; First posted 2019-06-03 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Depressive Symptoms
Keywords: breast cancer; mindfulness based intervention; cognitive behavioral therapy; depressive symptoms
MeSH Terms: conditions — Breast Neoplasms; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Intervention (Experimental): 8 group sessions lasting 2.5 hours each, on a weekly basis.
  Interventions: Behavioral: Mindfulness Based Intervention
- Cognitive Behavioral Therapy (Active Comparator): 8 group sessions lasting 2.5 hours each, on a weekly basis.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention — The MBI used in this study is called body-affective mindfulness (BAM); BAM is based on:
  (1) awareness practices such as body scan, breath meditation, walking meditation and yoga exercises; (2) mindfulness in relationship practices such as loving kindness, enriching listening to nature and persons and self-compassion; (3) sensorimotor psychotherapy Sensorimotor psychotherapy emphasizes the use of somatic resources to attain and sustain a mindful disposition and integrates the concept of a stress response with the concept of a "window of tolerance" in order to maximize the clinical utility of the intervention and tailor it to breast cancer patients.
  Other Names: MBI; BAM
  Arms: Mindfulness Based Intervention
Behavioral: Cognitive Behavioral Therapy — Cognitive behavior therapies will include cognitive restructuring, relaxation, skills training, and visual imagery, among other modalities.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Breast cancer is the most common cancer pathology among women worldwide and represents a complex psychological challenge for those affected. Diagnosis and subsequent treatments can have a significant impact not only on the physical well-being of people, but also on their psychological well-being. Tumor-related distress is described as an "unpleasant emotional multifactorial experience of a psychological, social and / or spiritual nature that can interfere with the ability to effectively cope with cancer, physical symptoms and treatment" from the National Comprehensive Cancer Network.Studies have shown that from one third to half of breast cancer patients can experience psychological distress. The psychological distress, understood as symptoms of anxiety, depression and stress, is related to a lower quality of life, a lower compliance related to a lower efficacy of the treatments, a higher mortality and a higher risk of suicide, so much so that this discomfort it is recognized as the sixth vital sign in cancer treatment. Both the diagnosis of cancer and the treatments related to the disease, can lead to the alternation of depressive phases and in some cases even to the presence of major depression: it is estimated that the levels of depression reach thresholds that oscillate between 5 and 25% between women suffering from breast cancer.

In reference to what are the interventions aimed at reducing depressive symptomatology in patients with breast cancer, in this study we refer in particular to 2 treatments, of which several studies attest to their effectiveness: interventions based on Mindfulness (MBI) and interventions based on cognitive behavioral therapy (CBT).

Cognitive-behavioral therapy (CBT) is an empirically supported treatment for depression. Numerous studies have shown that CBT is both effective in treating acute depression and preventing subsequent relapses and relapses after the end of active treatment.

MBI-based interventions have been widely disseminated both at the clinical and research level as short, cost-effective interventions.

Several systematic reviews have shown the effectiveness of MBIs in improving anxiety and depressive symptoms, sleep, fatigue, disease adaptation and stress reduction, with coping and well-being improved in patients with chronic illnesses including also the oncological pathologies. In particular, a meta-analysis of studies conducted on women with breast cancer confirmed the effectiveness of MBI in reducing symptoms of anxiety, depression and stress, suggesting the importance of these treatments in improving the mental health of these women. In addition, studies have shown that the improvements achieved are stable even at long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer;
* understanding of the Italian language;
* interruption of all psychotropic drugs at least one month before treatment and maintenance of interruption throughout the study or maintenance at baseline level;
* legal capacity to express consent to the processing;
* completion of all treatments except hormone therapy or trastuzumab at least 1 month before;
* score> of 13 and <of 30 at the BDI (Beck Depression Inventory (BDI);
* the ability to use at least e-mail management applications.

Exclusion Criteria:

* presence of serious psychological or psychiatric disorder, (eg severe major depressive disorder, psychotic disorder and bipolar disorder or abuse of active substances);
* severe suicidal tendency;
* presence of overt dementia;
* previous participation in groups of Mindfulness Based Intervention and Cognitive Behavioral Therapy groups.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in depression symptoms | week 0, week 8, week 20, week 44
  Beck Depression Inventory (BDI)
changes in depression and anxiety symptoms | week 0, week 8, week 20, week 44
  Depression Anxiety Stress Scale
changes in HRV | week 0, week 8, week 20, week 44
  Heart Rate Variability evaluation during practice

SECONDARY OUTCOMES:
changes in brest cancer quality of life | week 0, week 8, week 20, week 44
  Functional Assessment of Cancer Therapy - Breast (FACT-B)
changes in fatigue | week 0, week 8, week 20, week 44
  Additional Concern Subscale of the Functional Assessment of Illness Therapy - Fatigue subscale (FACIT-F)
changes in self compassion | week 0, week 8, week 20, week 44
  Self-Compassion Scale-forma breve (SCS-SF)
changes in sleep quality | week 0, week 8, week 20, week 44
  Pittsburgh Sleep Quality Index (PSQI)
changes in attention and self awareness | week 0, week 8, week 20, week 44
  Mindfulness Awareness Attention Scale (MAAS)
changes in trauma sypmtoms | week 0, week 8, week 20, week 44
  Impact of Event Scale - Revised (IES-R)

IPD SHARING:
Plan to Share IPD: Undecided